CLINICAL TRIAL: NCT06307665
Title: A Randomized, Double-blind, Multicenter, Parallel-group, Phase IIIb 52 Week Study Evaluating the Efficacy and Safety of PT027 Compared With PT007 Administered as Needed in Participants 12 to < 18 Years of Age With Asthma (ACADIA)
Brief Title: Evaluating the Efficacy and Safety of PT027 Compared With PT007 Administered As Needed in Participants 12 to < 18 Years of Age With Asthma
Acronym: ACADIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6934C00001
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Fast-acting β2-agonist; Metered-Dose Inhaler (MDI); Bronchodilatory; Inhaled corticosteroids; Anti-inflammatory; Rescue Therapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Budesonide/albuterol metered -dose inhaler (BDA MDI) (Experimental): Participants will receive BDA MDI 160/180 μg (given as 2 puffs of 80/90 μg) as needed.
  Interventions: Combination Product: BDA MDI
- Albuterol sulfate metered-dose inhaler (AS MDI) (Active Comparator): Participants will receive AS MDI 180 μg (given as 2 puffs of 90 μg) as needed.
  Interventions: Combination Product: AS MDI

INTERVENTIONS:
Combination Product: BDA MDI — Participants will receive oral inhalation of BDA MDI 160/180 μg taken as 2 puffs of 80/90 μg as needed.
  Other Names: PT027
  Arms: Budesonide/albuterol metered -dose inhaler (BDA MDI)
Combination Product: AS MDI — Participants will receive oral inhalation of AS MDI 180 μg taken as 2 puffs of 90 μg as needed.
  Other Names: PT007
  Arms: Albuterol sulfate metered-dose inhaler (AS MDI)

SUMMARY:
The purpose of this study is to compare the effect of budesonide/albuterol metered-dose inhaler (BDA MDI) with albuterol sulfate metered-dose inhaler (AS MDI), both administered as needed, on the annualized rate of severe asthma exacerbations in adolescents with a documented clinical diagnosis of asthma and at least one severe exacerbation in the prior year.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multicenter, parallel-group Phase IIIb study with a fixed treatment period of 52 weeks.

The study will consist of 3 periods:

1. Screening period (7 to 28 days)
2. Treatment period of 52 weeks
3. Safety follow-up period (7 to 14 days after the end of treatment [EOT] visit)

Participants who meet the eligibility criteria will be randomly assigned to BDA MDI 160/180 micrograms (μg) or AS MDI 180 μg treatment groups in a 1:1 ratio on top of their own usual maintenance therapy during treatment period.

This study will also include a pharmacokinetic (PK) sub-study with single visit scheduled after the safety follow-up visit in the main study. During PK sub-study, single dose of open-label BDA MDI 160/180 μg will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of asthma at least 12 months.
* Receiving one of the following scheduled asthma maintenance therapies for at least 3 months with stable dosing for at least the last one month

  1. Low-to-high-dose Inhaled corticosteroid(s) (ICS)
  2. Low-to-high-dose ICS or ICS/long-acting β2-agonist (LABA) with or without one additional maintenance therapy from the following: leukotriene receptor antagonist (LTRA), long-acting muscarinic antagonist (LAMA), or theophylline
* Receiving inhaled short-acting β2-agonist (SABA) as needed.
* A documented history of at least one severe asthma exacerbation within 12 months.
* Use of Sponsor-provided albuterol sulfate inhalation aerosol medication.
* Demonstrate acceptable MDI administration technique as assessed by the investigator; use of spacers is prohibited.
* Able to perform acceptable and reproducible peak expiratory flow (PEF) measurements as assessed by the investigator.
* Participants must adhere to protocol specific contraception methods.
* Negative urine pregnancy test for participants of childbearing potential.
* Have a BMI < 40 kg/ m^2.
* Capable of giving assent (signing the assent form) to participate in the study which includes compliance with the requirements and restrictions. The caregiver of the patient must be capable of giving written informed consent for the patient's participation in the study. Consent and assent forms must be completed prior to any study-specific procedures.

Exclusion Criteria:

* Life-threatening asthma defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s).
* Experienced > 3 severe asthma exacerbations within 12 months before screening.
* Completed treatment for lower respiratory infection and severe asthma exacerbation with SCS within 4 weeks of screening.
* Upper respiratory infection involving antibiotic treatment not resolved.
* Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months (including all forms of tobacco, e-cigarettes [vaping], and marijuana).
* Other significant lung disease, including regular or occasional use of oxygen.
* Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, hematological, neuropsychological, endocrine, or gastrointestinal disorders.
* Cancer not in complete remission for at least 5 years.
* History or hospitalization for psychiatric disorder or attempted suicide within one year.
* Significant abuse of alcohol or drugs, in the opinion of the investigator.
* Oral corticosteroid(s) (OCS)/SCS use (any dose and any indication) within 4 weeks before Visit 1 or chronic use of OCS/SCS (≥ 3 weeks use in 3 months prior to Visit 1).
* Use of any oral SABAs within one month.
* Having a known or suspected hypersensitivity to albuterol/salbutamol, or budesonide and/or their excipients.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-10-13 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of severe asthma exacerbations (AAER) | From Randomization (Day 1) to Week 52 (EOT)
  The effect of BDA MDI compared with AS MDI, both administered as needed, on the AAER in participants with asthma will be evaluated.

SECONDARY OUTCOMES:
Time to first (TTF) severe asthma exacerbation | From Randomization (Day 1) to Week 52 (EOT)
  The effect of BDA MDI compared with AS MDI, both administered as needed, on the risk of a first severe asthma exacerbation in participants with asthma will be evaluated.
Annualized total systemic corticosteroids (SCS) exposure for treatment of asthma | From Randomization (Day 1) to Week 52 (EOT)
  The effect of BDA MDI compared with AS MDI, both administered as needed, on the annualized total SCS exposure for treatment of asthma in participants with asthma will be evaluated.
Number of participants with adverse events (AEs) and severe adverse events (SAEs) | Up to Week 52
  The safety and tolerability of BDA MDI compared with AS MDI in participants with asthma will be assessed.
Maximum Observed Concentration (Cmax) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Area under concentration-time curve from time 0 to last quantifiable concentration (AUClast) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Area under concentration-time curve from time 0 to infinity (AUCinf) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Time to reach maximum concentration following drug administration (Tmax) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Time of last quantifiable concentration (Tlast) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Terminal elimination half-life (t½λz) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Terminal elimination rate constant (λz) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Apparent total body clearance (CL/F) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.
Apparent volume of distribution based on the terminal phase (Vz/F) | At 0, 10, 20, 40 minutes and 1, 2, 4, 6, 8, 10, and 12 hours post-dose
  The PK of budesonide and albuterol in participants with asthma, following a single dose of BDA MDI will be characterized.

CONTACTS AND LOCATIONS:
Locations (111):
- United States (86):
  - Research Site, Anchorage, Alaska
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Long Beach, California
  - Research Site, Madera, California
  - Research Site, Mission Viejo, California
  - Research Site, Moreno Valley, California
  - Research Site, Orange, California
  - Research Site, Riverside, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Westminster, California
  - Research Site, Denver, Colorado
  - Research Site, Wilmington, Delaware
  - Research Site, Destin, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Fayetteville, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Normal, Illinois
  - Research Site, River Forest, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Lafayette, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Ellicott City, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Mankato, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Newark, New Jersey
  - Research Site, Northfield, New Jersey
  - Research Site, Ocean City, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Cortland, New York
  - Research Site, Hawthorne, New York
  - Research Site, Hollis, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Vestal, New York
  - Research Site, Watertown, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Findlay, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Yukon, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Baytown, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Bellaire, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, Frisco, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, McKinney, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Burke, Virginia
  - Research Site, Bellingham, Washington
  - Research Site, Vancouver, Washington
- China (16):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Hohhot
  - Research Site, Mianyang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Yanji
  - Research Site, Yantai
  - Research Site, Zhongshan
- Mexico (3):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Monterrey
- South Africa (6):
  - Research Site, Durban
  - Research Site, Krugersdorp
  - Research Site, Middelburg
  - Research Site, Panorama
  - Research Site, Somerset West
  - Research Site, Welkom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/